CLINICAL TRIAL: NCT01071655
Title: Selecting Treatment in Colorectal Cancer: Capecitabine or 5-fluorouracil Selection According to Polymorphisms in TS-3'UTR and ERCC1-118 to be Combined With Oxaliplatin or Irinotecan as First-line Chemotherapy in Advanced Colorectal Cancer
Brief Title: Selecting Treatment in Colorectal Cancer:Capecitabine or 5-fluorouracil Selection to be Combined With Oxaliplatin or Irinotecan as First-line Chemotherapy in Advanced Colorectal Cancer
Acronym: SETICC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTD-09-01(ML25052); 2009-012562-31 (EudraCT Number)
Record Dates: First submitted 2010-02-15; First posted 2010-02-19 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; Bevacizumab; Oxaliplatin; Irinotecan; 5FU; capecitabine
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): Patients with zero favorable genotype: BVZ + XELIRI.
  Patients with one favorable genotype: TS 3'UTR +6bp/+6bp and ERCC1-118 T/T: BVZ + XELOX or TS 3'UTR +6bp/-6bp and ERCC1-118 C/T ó C/C: BVZ + FUIRI.
  Patients with two favorable genotypes : BVZ + FUOX.
  Interventions: Drug: BVZ+XELOX or BVZ+XELIRI or BVZ+FUIRI or BVZ+FUOX
- 1 (Active Comparator): BVZ + XELOX
  Interventions: Drug: BVZ+XELOX

INTERVENTIONS:
Drug: BVZ+XELOX or BVZ+XELIRI or BVZ+FUIRI or BVZ+FUOX — BVZ + XELOX. Bevacizumab 7,5 mg/kg day 1; capecitabine 1000 mg/m2/12 h days 1-14; oxaliplatin 130 mg/m2 day 1
  BVZ + XELIRI. Bevacizumab 7,5 mg/kg day 1; Capecitabine 800 mg/m2/12 h days 1-14; Irinotecan 200 mg/m2 day 1
  BVZ + FUIRI. Bevacizumab 5 mg/kg biweekly; 5-FU 2.250 mg/m2 weekly; Irinotecan 80 mg/m2 weekly
  BVZ + FUOX. Bevacizumab 5 mg/kg biweekly; 5-FU 2.250 mg/m2 weekly; Oxaliplatin 85 mg/m2 biweekly
  Arms: 2
Drug: BVZ+XELOX — BVZ + XELOX. Bevacizumab 7,5 mg/kg day 1; capecitabine 1000 mg/m2/12 h days 1-14; oxaliplatin 130 mg/m2 day 1
  Arms: 1

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of the capecitabine or 5-fluorouracil selection, according to polymorphisms in TS-3'UTR and ERCC1-118, to be combined with oxaliplatin or irinotecan as first-line chemotherapy in advanced colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* informed consent signed
* Histological or citological adenocarcinoma confirmation carcinoma on the colon or colorectal metastatic or relapsed patients with adenocarcinoma of colon or recto, confirmed histologically with metastatic disease
* measurable disease (following RECIST criteria)
* ECOG ≤ 2
* older or equal 18 years old
* life expectancy superior to 3 months
* Adequate or moderate renal function: renal function (Creatinine clearance > 30mL/min), based on Cockroff - Gault.
* Potential fertile women negative pregnancy test in serum or urine, 10 days prior the first study dose given
* Use an adequate contraceptive method

Exclusion Criteria:

* Patients treated previously with Bevacizumab
* Non measurable lesion as only disease evidence
* Previous chemotherapy treatment for adjuvant or neoadjuvant disease (no metastatic (M0), or immunotherapy active/passive for the advance or metastatic disease. It is permitted the adjuvant or neoadjuvant treatment it is has finished at least 6 months before the initiation of the study drug.If the patient has received an adjuvant treatment previously the patient cannot participate if disease progression has been confirmed during the treatment or on the 6 months later
* Prior radiotherapy is allowed if it has not been administered in the target lesions selected for this study, unless progression of said lesions in the irradiated field is documented, and as long as treatment has concluded at least 4 weeks before beginning the study.
* Prior surgical treatment of the disease in stage IV is allowed
* Functional dependency
* Previous serious adverse events or unexpected to fluoropyrimidine treatment and /o patients with proved deficit in dehidropirimidin dehydrogenase (DPD)
* Patients classified as "weak or fragile"
* Cardiac concomitant present: Symptomatic auriculoventricular arrhythmia history, and / cardiac arrhythmias requiring medication or peripheral vascular disease, grade II or higher. Furthermore, those patients who have had a myocardial infarction in the year prior to beginning the treatment of the study will be excluded.
* History of another neoplastic disease during the last five years, with the exception of cured basal cell carcinoma of the skin and cervical carcinoma in situ.
* History or indications of CNS disease in the physical examination.
* History of psychiatric disability that the investigator considers clinically significant, which prevents the patient from granting the informed consent or interferes with compliance of taking the oral medication.
* Uncontrolled hypertension or clinically significant (i.e. active) cardiovascular disease: CVA/stoke (≤ 6 months prior to randomisation), myocardial infarction (≤ 6 months prior to randomisation), unstable angina, New York Heart Association (NYHA,) Grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome or inability to take oral medication.
* Patients subjected to organ allograft who require immunosuppressive treatment.
* Severe, non-cicatrized osseous fractures, wounds or ulcers
* Indications of hemorrhagic diathesis or coagulopathy.
* Severe, uncontrolled intercurrent infections or other severe, uncontrolled concomitant diseases.
* Any of the following laboratory values:

  1. Absolute neutrophil count (ANC) < 1.5 x 109/l
  2. Platelet count < 100 x 109/l
  3. Hemoglobin < 10 g/dl (it can be transfused to maintain or exceed this level)
  4. International Normalized Ratio (INR) > 1.5
  5. Total bilirubin > 1.5 times the upper limit of normal (ULN)
  6. ALAT, ASAT > 2.5 x ULN or > 5 x (ULN) in the case of hepatic metastases
  7. Alkaline phosphatase > 2.5 x ULN or > 5 x ULN in the case of hepatic metastases or > 10 x ULN in the case of osseous metastases.
* Patients subjected to a major surgical procedure, open biopsy or who have had significant traumatic lesions within the 28 days prior to beginning the treatment of the study or in whom it is foreseen that a major surgical procedure will be necessary during the course of the study; fine-needle aspiration within the 7 days prior to beginning the treatment of the study.
* Current or recent use (within the 10 days prior to beginning the treatment of the study) of oral or parenteral anticoagulants at complete doses or thrombolytic agents. The use of low doses of warfarin is allowed, with an International Normalized Ratio [INR] of < 1.5.
* Daily chronic treatment with high doses of aspirin (> 325 mg/day) or non-steroid anti-inflammatory medications (which inhibit the platelet function at doses used for treating chronic inflammatory diseases).
* Patients who have received any drug or agent/procedure under research, i.e., who have participated in another clinical trial during the 4 weeks prior to beginning the treatment with the medications of the study.
* Pregnancy or lactating woman. Woman with reproductive potential unless using an effective method of contraception (Postmenopausal woman must have been amenorrheic during at least 12 months).
* Known hypersensitivity to any of the study drugs or excipients of the Bevacizumab or to Chinese hamster ovary cell products or to other recombinant human or humanised antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2010-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 2010-2014

SECONDARY OUTCOMES:
overall survival | 2010-2014
Objective response rate | 2010-2014
% of patients whose disease becomes resectable | 2010-2014
Adverse events | 2010-2014
Evaluation of KRAS status as a molecular marker | 2010-2014

CONTACTS AND LOCATIONS:
Overall Officials: Albert Abad, Study Chair — Institut Català d'Oncologia.Hospital Universitari Germans Trias i Pujol. Badalona. Spain
Locations (1):
- Spanish Cooperative Group for Gastrointestinal Tumour Therapy, Madrid, Spain

REFERENCES:
- [Derived] Abad A, Martinez-Balibrea E, Vieitez JM, Alonso-Orduna V, Garcia Alfonso P, Manzano JL, Massuti B, Benavides M, Carrato A, Zanui M, Gallego J, Gravalos C, Conde V, Provencio M, Valladares-Ayerbes M, Salazar R, Sastre J, Montagut C, Rivera F, Aranda E. Genotype-based selection of treatment of patients with advanced colorectal cancer (SETICC): a pharmacogenetic-based randomized phase II trial. Ann Oncol. 2018 Feb 1;29(2):439-444. doi: 10.1093/annonc/mdx737. PMID 29145602
- See also: Related Info — http://www.ttdgroup.org